CLINICAL TRIAL: NCT01302457
Title: Oral Care Study on Burn Patients
Status: Withdrawn | Type: Observational
Sponsor: Saint Elizabeth Regional Medical Center (Other)
Responsible Party: Saint Elizabeth Regional Medical Center, Saint Elizabeth Regional Medical Center
Other Study IDs: 609-036
Record Dates: First submitted 2011-02-09; First posted 2011-02-24 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Burn
Keywords: Thermal Burn Trauma
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Same Subjects: The control group will be 19 years or older and be randomly picked from from volunteer staff at Saint Elizabeth Regional Medical Center. This is a prospective study that will look at the similarities and difference of both groups. This will help us determine if there is a need to improve oral hygiene protocol given to burn/intensive care patients. Each group will consist of 25 subjects
- Health Volunteers: The control group will be 19 years or older and be randomly picked from volunteer staff at Saint Elizabeth Regional Medical Center.
  DESIGN This is a prospective study that will look at the similarities and difference of both groups. This will help us determine if there is a need to improve oral hygiene protocol given to burn/intensive care patients. Each group will consist of 25 subjects

SUMMARY:
There have been multiple articles done regarding oral hygiene on patients in burn and intensive care patients. All articles agree the need for good oral hygiene in these special needs patients. They also note that more research needs to be done on this subject, yet have no direction of how to proceed in this research. Currently, no research has been done on the burn/intensive care patient to see if there is a difference form the non-hospitalized patient which oral hygiene protocol is based on.

DETAILED DESCRIPTION:
BACKGROUND IMFORATION AND INTRODUCTION There have been multiple articles done regarding oral hygiene on patients in burn and intensive care patients. All articles agree the need for good oral hygiene in these special needs patients. They also note that more research needs to be done on this subject, yet have no direction of how to proceed in this research. Currently, no research has been done on the burn/intensive care patient to see if there is a difference form the non-hospitalized patient which oral hygiene protocol is based on.

OJECTIVE The primary purpose of this prospective study is to determine if the burn/intensive care patient's oral condition is similar or different from the normal standard.

PATIENT SELECTION CRITERIA

1. Patients age must be 19 and older.
2. Patients must be on a ventilator in the burn or intensive care unit.
3. The control group will be 19 years or older and be randomly picked from from volunteer staff at Saint Elizabeth Regional Medical Center.

DESIGN This is a prospective study that will look at the similarities and difference of both groups. This will help us determine if there is a need to improve oral hygiene protocol given to burn/intensive care patients. Each group will consist of 25 subjects

ELIGIBILITY:
Inclusion Criteria:PATIENT SELECTION CRITERIA

1. Patients age must be 19 and older.
2. Patients must be on a ventilator in the burn or intensive care unit.
3. The control group of Healthy Volunteers will be 19 years or older and be randomly picked from volunteer staff at Saint Elizabeth Regional Medical Center.

Exclusion Criteria:

* Unable to complete Informed Consent Process

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PATIENT SELECTION CRITERIA
  1. Patients age must be 19 and older.
  2. Patients must be on a ventilator in the burn or intensive care unit.
  3. The control group will be 19 years or older and be randomly picked from volunteer staff at Saint Elizabeth Regional Medical Center.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Patient's Oral Condition | 30 days
  The primary purpose of this prospective study is to determine if the burn/intensive care patient's oral condition is similar or different from the normal standard.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Burgess, D.D.S., Principal Investigator — Saint Elizabeth Regional Medical Center
Locations (1):
- Saint Elizabeth Regional Medical Center, Lincoln, Nebraska, United States